CLINICAL TRIAL: NCT02431988
Title: COBALT: Evaluation of CAR19 T-cells as an Optimal Bridge to Allogeneic Transplantation
Brief Title: Evaluation of CAR19 T-cells as an Optimal Bridge to Allogeneic Transplantation
Acronym: COBALT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/14/0385; 2015-000348-40 (EudraCT Number)
Record Dates: First submitted 2015-03-23; First posted 2015-05-01 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Relapsed; refractory; DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — Leukapheresis; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR19 T-cells (Experimental): Patients will receive a single infusion of CAR19 T-cells following standard pre-conditioning with cyclophosphamide and fludarabine.
  The CAR19 T-cells are to be administered on day 0.
  Interventions: Procedure: Leukapheresis; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: CAR19 T-Cells

INTERVENTIONS:
Procedure: Leukapheresis — Patients will undergo leukapheresis prior to pre-conditioning chemotherapy to provide the immune cells required to produce the therapeutic product.
Drug: Cyclophosphamide — Patients will receive a standard pre-conditioning regime with cyclophosphamide 60mg/kg/day IV over 1 hour for 2 days (day-7 and day-6).
Drug: Fludarabine — Fludarabine 25mg/m2/day IV over 15/30 minutes for 5 days (Day-5 to day-1).
Biological: CAR19 T-Cells — The CAR19 T-cells are to be administered on day 0 at the dose specified by the Cancer Trials Centre (CTC) at the time of registration.
  Three dose cohorts are planned:
  * Dose Level 1: 2x105 CAR19 T-cells/kg
  * Dose Level 2: 1x106 CAR19 T-cells/kg
  * Dose Level 3: 5x106 CAR19 T-cells/kg
  Other Names: CD19 specific Chimeric Antigen Receptor T-cells

SUMMARY:
The purpose of this study is to administer novel cluster of differentiation antigen 19 (CD19) specific Chimeric Antigen Receptor T-cells (CAR19 T-cells) to patients with relapsed or resistant Diffuse Large B Cell Lymphoma (DLBCL) to assess the safety and efficacy of this strategy as a bridge to allogeneic transplantation.

DETAILED DESCRIPTION:
Patients with Diffuse Large B Cell Lymphoma (DLBCL) resistant to or relapsing following rituximab-containing chemotherapy regimens have a poor prognosis. Patients may receive salvage chemotherapy and possibly an autologous stem cell transplant (auto-SCT). A proportion of these patients, however, will not respond to the chemotherapy or may relapse after the auto-SCT and therefore require novel treatment options. Such patients may benefit from an allogeneic stem cell transplantation (allo-STC).

In this study the investigators aim to administer CAR19 T-cells to act as a bridge to the transplant strategy. Specifically, (1) the feasibility of generating CD19 specific Chimeric Antigen Receptor T-cells called CAR19 T-cells, (2) the safety of administering the CD19 CAR T-cells in this setting, (3) how well the CAR19 T-cells engraft and (4) to evaluate how effective these cells are as a bridge to allogeneic transplantation.

Following informed consent and registration to the trial, patients will undergo an unstimulated leucapheresis for generation of the CAR19 T cells. Whilst the cells are being generated, patients will proceed with a further cycle of standard salvage (recommended ifosfamide, epirubicin and etoposide (i.e. the IVE regime), and should not receive rituximab. Patients will receive pre-conditioning with intravenous fludarabine and cyclophosphamide prior to infusion of a single dose of CAR-modified T-cells. An escalating dose protocol will be employed to identify a minimum effective dose of CAR19 T-cells.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-65 years
2. Confirmed diagnosis of CD19+ DLBCL
3. Primary resistant or relapsed disease failing to achieve metabolic Complete Response (CR) to 1st line salvage, or relapse post autograft failing to achieve metabolic CR following a single further cycle of salvage
4. Potential allogeneic transplant candidate
5. Agreement to have a pregnancy test, use adequate contraception for 12 months post-CAR19 T-cell infusion
6. Karnofsky performance status >60
7. Written informed consent

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Prior allogeneic transplantation
3. Progressive disease following most recent salvage prior to planned leucapheresis (those with mixed response are eligible)
4. Prior history of ischaemic heart disease, dysrhythmias, abnormal electrocardiogram (ECG)(Left Bundle Branch Block (LBBB)), Multiple Gated Acquisition (MUGA) left ventricular ejection fraction (LVEF) <40%
5. Exclusions for proceeding to allogeneic transplantation (active hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV); liver function test (LFT) >3 x upper limit of normal (ULN); Creatinine Clearance (CrCl) <40 ml/min; or other comorbidity that precludes transplantation)
6. Known central nervous system (CNS) involvement or cerebral vascular accident (CVA) within prior 3 months
7. Patients receiving corticosteroids at a dose of > 10mg prednisolone per day (or equivalent)
8. Use of rituximab within the last 2 months prior to CAR19 T-cell infusion
9. Active autoimmune disease requiring immunosuppression
10. Life expectancy <3 months
11. Known allergy to albumin or dimethylsulfoxide (DMSO)
12. Any contraindication to the administration and use of ifosfamide, epirubicin, etoposide, fludarabine and cyclophosphamide.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of adequate leucapheresis collection and generation of CAR19 T cells. | 1 month
  The number of CAR19 T cells successfully manufactured as a fraction of the number of patients undergoing leukapheresis (all patients registered).
Toxicity evaluation following CAR19 T-cell administration. | 1 year
  Toxicity will be examined for each patient receiving CAR19 T cells, using the maximum grade for each toxicity type, all summarized as number of patients with adverse events.
Efficacy of CAR19 T-cells. | 1 year
  Efficacy will be defined as the number of patients that meet the clinical complete responders criteria.

SECONDARY OUTCOMES:
CAR19 T-cell engraftment | 1 year
  1. Engraftment, expansion and persistence of CAR19 T-cells. Detection of any level of CAR19 expression in circulating T cells (ie PBMC) by quantitative polymerase chain reaction (qPCR) and flow cytometry following infusion.
B cell compartment | 1 year
  2. Depletion of B cell compartment. The percentage reduction from baseline. Absolute B cell numbers measured by flow of PBMC (cells/ul) .
Cytokine profile | 1 year
  3. Timing and magnitude of cytokine release. Data on timing (kinetic of change) as the mean (or median) amount of cytokine (pg/ml) over a number of days post-infusion. Using the individual patient data, the mean (or median) time to peak value can be obtained.
  Magnitude - kinetic and peak of cytokine levels, notably Tumour Necrosis Factor-alpha (TNF-a), Interleukin- 6 (IL-6) and Interferon-gamma (IFN-g) (pg/ml), can be plotted for each patient, as means (or medians).
Clinical complete response | 1 month
  4. Clinical response evaluated using standard PET-CT criteria at day 28 compared to baseline scan. Proportion of patients with complete response will be calculated.
Eligibility to allogeneic transplantation | 1-3 years
  5. Number of patients proceeding to allogeneic transplantation out of all patients registered to the trial, and also only for those who received CAR19 T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Peggs, Study Chair — University College, London
Locations (1):
- University College London Hospital, London, United Kingdom

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338